CLINICAL TRIAL: NCT05040776
Title: Prospective, Open-Label Single Ascending Dose Study of Two Dose Levels of Frunexian (EP-7041), Followed by a Randomized Comparison of One Dose With Institutional Standard Care, for Thromboprophylaxis in Patients Managed in Intensive Care Settings for COVID-19 Syndrome: The COVID-ThromboprophylaXIs Study
Brief Title: COVID-19 ThromboprophylaXIs Study of Novel FXIa Inhibitor Frunexian (EP-7041) in ICU Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: eXIthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-eXIthera-Prophy-001
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Thrombopenia; Covid19
MeSH Terms: conditions — Thrombocytopenia; COVID-19 | interventions — (2S,3R)-3-((2-aminopyridin-4-yl)methyl)-1-(((1R)-1-cyclohexylethyl) carbamoyl)-4-oxoazetidine-2-carboxylic acid

STUDY DESIGN:
Intervention Model Description: Multicenter, Open Label, Single Dose Escalation Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Other): Frunexian infusion 0.6 mg/kg/hr or 1 mg/kg/hr. 0.6 mg/kg/hr dose will be completed first.
  Interventions: Drug: EP-7041 Injection
- Institutional Standard (Active Comparator): Clinician's choice of prophylaxis strategy
  Interventions: Drug: EP-7041 Injection

INTERVENTIONS:
Drug: EP-7041 Injection — EP-7041 infusion
  Other Names: EP-7041; Frunexian

SUMMARY:
This is a multicenter, open-label, single cohort study of patients with confirmed COVID-19 syndrome who based on clinical judgment require care in an intensive care unit, regardless of whether or not mechanical ventilation is in use or is anticipated. Patients should be enrolled on the first day of the ICU stay; withdrawal of prior thromboprophylaxis, if any, will follow specific protocol guidance. Enrolled patients will thereafter be administered intravenous frunexian (EP-7041) until disposition from the hospital (including post-ICU non-critical care management)

DETAILED DESCRIPTION:
The goal of the COVID-ThromboprophylaXIs Study is to determine the safety and tolerability of two doses of frunexian (EP-7041) for the prevention of thromboembolism in the management of COVID-19 patients, compared to control patients managed with institutional standard care thromboprophylaxis regimens. Dosing of frunexian for the first 15 patients enrolled will be randomized to 0.6 mg/kg/hr IV (n=15) and next 15 patients will be randomized to 1.0 mg/kg/hr IV (n=15) for the duration of the index hospitalization. Enrollment will be paused after treatment of these 30 patients, at which time a dedicated DSMB will evaluate all collected safety data through 7 days post-index hospital discharge. If no adverse safety signal is identified for the 1.0 mg/kg/hr dose, enrollment will be resumed with the study dose of frunexian randomized 2:1 to 1.0 mg/kg/hr or institutional standard care for thromboprophylaxis in ICU patients with COVID-19. If safety concerns are identified for the higher dose and not for the lower dose, then open-label randomized enrollment vs institutional standard of care for thromboprophylaxis will proceed with an frunexian dose of 0.6 mg/kg/hr. The second phase of the study will enroll 60 additional patients, with 40 in the frunexian dosing arm, and 20 in the standard care arm.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 test (by local evaluation) positive
* Symptom severity and general risk of decompensation warrants, in the opinion of the treating clinician, admission to/care in an intensive care unit setting
* Patient or legally authorized representative (LAR) able and willing to provide written informed consent
* No contraindication to receiving anticoagulation
* At least one D-dimer value ≥2 times local ULN (within 72 hours of hospital admission)

Exclusion criteria

Patients who meet ANY of the following criteria are not eligible for inclusion:

* Moribund patient not expected to survive 24 hours
* ICU length of stay > 24 hours prior to initiation of frunexian infusion
* Existing venous thromboembolism
* Known immune compromise (HIV/AIDS, chemotherapy, chronic corticosteroid therapy, transplant patient, etc.)
* Active cancer diagnosis
* Pregnant, lactating, or parturient woman
* bodyweight <40kg
* hemoglobin <8.0 g/L in the last 72 hours
* platelet count <50 x 109/L in the last 72 hours
* known fibrinogen <1.5 g/L (if testing deemed clinically indicated by the treating physician prior to the initiation of anticoagulation)
* known INR >1.8 (if testing deemed clinically indicated by the treating physician prior to the initiation of anticoagulation)
* patient already on therapeutic anticoagulation at the time of screening (low or high dose nomogram UFH, LMWH, warfarin, or any regular dose of a direct oral anticoagulant)
* patient on dual antiplatelet therapy, when at least one of the agents cannot be stopped safely
* history of spontaneous intracranial bleeding; gastrointestinal bleeding requiring hospitalization and/or transfusion within prior 3 months
* major surgery within prior 30 days
* known bleeding within the last 30 days requiring emergency department presentation or hospitalization
* known history of a bleeding disorder of an inherited or active acquired bleeding disorder
* recent (<48 hours) or planned spinal or epidural anesthesia or puncture
* anticipated transfer to another hospital that is not a study site within 72 hours
* enrollment in other trials related to anticoagulation or antiplatelet therapy
* use of pneumatic compression devices for thromboprophylaxis
* Failure to meet ALL Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days after discharge
  Identify the appropriate dose of EP-7041 that demonstrates safety as defined by incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Charles V. Pollack, Jr.,, MA, MD, Study Director — Department of Emergency Medicine, University of Mississippi School of Medicine
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No